CLINICAL TRIAL: NCT01890876
Title: Altitude-dependent Effects of Concentric and Eccentric Exercise on Glucose Metabolism in Pre-diabetic Men
Brief Title: Altitude, Exercise and Glucose Metabolism in Pre-diabetic Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaet Innsbruck (Other)
Collaborators: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Martin Burtscher, Univ.-Prof. Mag. DDr. Martin Burtscher, Universitaet Innsbruck
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AN5029
Record Dates: First submitted 2013-06-27; First posted 2013-07-02 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Diabetes
Keywords: glucose tolerance, hypoxia, myokines, exercise
MeSH Terms: conditions — Diabetes Mellitus; Hypoxia; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low altitude (Active Comparator): Walking uphill Walking downhill
  Interventions: Other: Walking uphill; Other: Walking downhill
- High altitude (Active Comparator): Walking uphill Walking downhill
  Interventions: Other: Walking uphill; Other: Walking downhill

INTERVENTIONS:
Other: Walking uphill — ascending about 500 m
Other: Walking downhill — descending about 500 m

SUMMARY:
Concentric (CE) and eccentric (EE) exercises may differently affect glucose metabolism which may be additionally modified when exercises are performed in hypoxia, e.g. at moderate (1500 - 2500 m) or high (2500 - 3500 m) altitudes. However, data on the effects of glucose metabolism due to CE and EE in hypoxia are scarce but would be of utmost importance considering the increasing number of persons suffering from impaired glucose tolerance or diabetes and the unique opportunities provided by the mountainous regions of the Alps to perform CE (e.g. uphill hiking) and EE (downhill hiking, downhill skiing) at altitude between 1500 - 3500 m. Metabolic responses to exercise may be largely mediated by interleukin 6 (IL-6), which is predominantly derived from the contracting limbs and may support the maintenance of metabolic homeostasis during exercise. In addition, IL-6 is elevated with acute and chronic altitude exposure at least partly mediated via adrenergic stimulation. Thus, the type of exercise as well as hypoxia may contribute to IL-6 elevations and differences in serum IL-6 concentrations might help to explain distinctions between responses of glucose metabolism to CE and EE at low and moderate to high altitude.

32 male subjects suffering from pre-diabetes will be randomly assigned to a downhill (EE) or uphill (CE) walking group performing 9 sessions at low altitude (860 - 1360 m) and 9 sessions at moderate to high altitude (2000 - 2500 m). Between normoxic and hypoxic condition will be a break of approximately 12 month. Measurements of glucose metabolism, IL-6 plasma concentration will be performed pre, mid (day 5) and post intervention. Moreover anthropometric, strength and exercise capacity characteristics will be performed pre and post intervention.

We hypothesize that EE in hypoxia is more effective in the modulation of glycemic control in pre-diabetic men than CE in hypoxia as well as EE and CE in normoxia. It is suggested that effects on glucose metabolism are associated with changes in plasma IL-6 concentrations. EE in hypoxia is expected to result in a more persistent rise of plasma IL-6 concentration than CE in hypoxia and in normoxia and to a more pronounced rise in plasma IL-6 than EE in normoxia.

DETAILED DESCRIPTION:
Not desired.

ELIGIBILITY:
Inclusion Criteria:

* Pre-diabetes
* male
* age 50-65 years

Exclusion Criteria:

* smoking
* BMI > 30 kg/m2
* diseases not compatible with intervention

Ages: 50 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Glucose tolerance | 18 months

SECONDARY OUTCOMES:
Myokines | 18 months
Cardiovascular fitness | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin Burtscher, Professor, Principal Investigator — department of sport science, medical section, university innsbruck
Locations (1):
- Department of Sport Science, Medical Section, University of Innsbruck, Innsbruck, Austria

REFERENCES:
- [Background] Drexel H, Saely CH, Langer P, Loruenser G, Marte T, Risch L, Hoefle G, Aczel S. Metabolic and anti-inflammatory benefits of eccentric endurance exercise - a pilot study. Eur J Clin Invest. 2008 Apr;38(4):218-26. doi: 10.1111/j.1365-2362.2008.01937.x. PMID 18339002
- [Background] Duennwald T, Gatterer H, Groop PH, Burtscher M, Bernardi L. Effects of a single bout of interval hypoxia on cardiorespiratory control and blood glucose in patients with type 2 diabetes. Diabetes Care. 2013 Aug;36(8):2183-9. doi: 10.2337/dc12-2113. Epub 2013 Mar 27. PMID 23536585
- [Background] Burtscher M, Gatterer H, Kunczicky H, Brandstatter E, Ulmer H. Supervised exercise in patients with impaired fasting glucose: impact on exercise capacity. Clin J Sport Med. 2009 Sep;19(5):394-8. doi: 10.1097/JSM.0b013e3181b8b6dc. PMID 19741312
- [Derived] Philippe M, Junker G, Gatterer H, Melmer A, Burtscher M. Acute effects of concentric and eccentric exercise matched for energy expenditure on glucose metabolism in healthy females: a randomized crossover trial. Springerplus. 2016 Aug 30;5(1):1455. doi: 10.1186/s40064-016-3062-z. eCollection 2016. PMID 27652031